CLINICAL TRIAL: NCT06883916
Title: Effect of Virtual Reality Environment Created in Preoperative Area and Hand Massage on Patient Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Nursevim Aydıngülü, Principal Investigator, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Faculty of Health Sciences
Record Dates: First submitted 2025-02-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Preoperative Patients; Surgical Procedures, Elective; Anxiety
Keywords: preoperative anxiety; preoperative patients; complementary and alternative therapies; massage; virtual reality
MeSH Terms: conditions — Anxiety Disorders | interventions — Massage

STUDY DESIGN:
Intervention Model Description: The study was conducted to investigate the effects of video watching with virtual reality glasses and classical hand massage on patient outcomes in patients undergoing elective surgery. It was planned as a three-group, randomized controlled and interventional study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality (Experimental): Patients in the preoperative waiting unit were shown a video using virtual reality glasses for 10 minutes.
  Interventions: Behavioral: Virtual reality tour
- Massage (Experimental): A hand massage lasting 5 minutes was applied to each hand by the researcher.
  Interventions: Behavioral: Massage

INTERVENTIONS:
Behavioral: Virtual reality tour — The glasses have a pre-loaded video containing nature images in their memory. The patient feels like they are walking in the natural environment shown in the video.
  Arms: Virtual Reality
Behavioral: Massage — A hand massage was applied by the researcher for 5 minutes for each hand. The massage, which was performed using baby oil and a paper towel, lasted 10 minutes in total for both hands.
  Arms: Massage

SUMMARY:
The aim of this study is to investigate the effects of video watching with virtual reality glasses and classical hand massage on patient outcomes in patients undergoing elective surgery. In addition, it's examined that if virtual reality glasses and hand massage execution is convenient way of to reduce anxiety in patients before surgery.

The main questions it aims to answer are:

* Is there a significant difference between the study groups in terms of post-application anxiety level?
* Is there a significant difference between the study groups in terms of post-application vital signs, pain and patient satisfaction? Researchers will compare responses to anxiety scales before and after the hand massage and virtual reality videos to see if they reduce anxiety levels.

Participants will:

* In the virtual reality group, they will answer the questions on the surgical anxiety scale, watch the video with VR glasses and answer the questions on the scale again.
* In the massage group, they will answer the questions on the surgical anxiety scale, and after the researcher gives them a hand massage, they will answer the questions on the scale again.

DETAILED DESCRIPTION:
Surgical Anxiety Scale: The scale was developed by Burton et al. in 2018 to assess preoperative anxiety levels. Each item of the 17-item scale is answered between 0 and 5 points. It consists of three sub-dimensions reflecting individuals' health status, recovery process, and anxiety about procedures. Health-related anxiety is calculated by adding the scores given to items 7, 8, 9, 10, 12, and 13; recovery-related anxiety is calculated by adding the scores given to items 2, 14, 16, and 17; and procedure-related anxiety is calculated by adding the scores given to items 1, 3, 4, and 5. The total score of the scale is calculated by adding the scores of all sub-dimensions and the scores of the three items not included in the sub-dimensions. A minimum of 0 and a maximum of 68 points can be obtained from the scale. Although there is no cut-off point for the scale, it can be said that surgical anxiety increases as the total score of the scale increases.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo elective surgery and whose general condition is ASA (American Society of Anesthesiology) classification I, II or III
* Patients who are not sedated
* Patients over the age of 18
* Patients without a psychiatric or behavioral diagnosis
* Patients who do not have a communication barrier due to hearing loss or spoken language

Exclusion Criteria:

* Vertigo and motion sickness
* Carpal tunnel syndrome
* Hand cuts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Surgical Anxiety Scale | The Surgical Anxiety Scale will be administered 5 minutes before the intervention assigned to the research groups (pre-test) and again 5 minutes after the completion of the massage or virtual reality intervention (post-test).
  The scale was developed by Burton et al. in 2018 to assess preoperative anxiety levels. Each item of the 17-item scale is answered between 0 and 5 points. It consists of three sub-dimensions reflecting individuals' health status, recovery process, and anxiety about procedures. Health-related anxiety is calculated by summing up items 7, 8, 9, 10, 12, and 13; recovery-related anxiety is calculated by summing up items 2, 14, 16, and 17; and procedure-related anxiety is calculated by summing up items 1, 3, 4, and 5. The total score of the scale is calculated by summing up all sub-dimension scores and the scores of three items not included in the sub-dimensions. A minimum of 0 and a maximum of 68 points can be obtained from the scale. A high total scale score indicates increased surgical anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Sevban A Professor doctor, Study Director — Cukurova University
Locations (1):
- Balcali Hospital Health Application and Research Center, Adana, Sarıçam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since the research is conducted with real persons, sharing personal data is not ethically appropriate.

REFERENCES:
- [Background] Bekelis K, Calnan D, Simmons N, MacKenzie TA, Kakoulides G. Effect of an Immersive Preoperative Virtual Reality Experience on Patient Reported Outcomes: A Randomized Controlled Trial. Ann Surg. 2017 Jun;265(6):1068-1073. doi: 10.1097/SLA.0000000000002094. PMID 27906757
- [Background] Niharika P, Reddy NV, Srujana P, Srikanth K, Daneswari V, Geetha KS. Effects of distraction using virtual reality technology on pain perception and anxiety levels in children during pulp therapy of primary molars. J Indian Soc Pedod Prev Dent. 2018 Oct-Dec;36(4):364-369. doi: 10.4103/JISPPD.JISPPD_1158_17. PMID 30324926
- See also: Effects of distraction using virtual reality technology on pain perception and anxiety levels in children during pulp therapy of primary molars — https://journals.lww.com/jped/fulltext/2018/36040/effects_of_distraction_using_virtual_reality.8.aspx
- Available data/document: Informed Consent Form: Ethics Committee Approval — https://tip.cu.edu.tr/storage/Mevzuat/Kurullar%20Y%C3%B6nergesi.pdf